CLINICAL TRIAL: NCT05690022
Title: The Use of EndoFlip as a Clinical Tool for the Prediction of Postoperative GERD After Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Clinical Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EndoFlip
Record Dates: First submitted 2022-12-13; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Gastroesophageal Reflux; Sleeve Gastrectomy; Bariatric Surgery Complication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Before/after study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Before sleeve gastrectomy (No Intervention): Gastroesophageal Reflux Disease (GERD) will be evaluated before surgery. EndoFlip, gastroscopy, pH-study and GERD-Health-Related Quality of Life Questionnaire will be realized for all patients.
- Sleeve gastrectomy (Experimental): After the surgical intervention, new onset or worsening of GERD will be evaluated.
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: sleeve gastrectomy — Patients will be recruited for a sleeve gastrectomy according to the guidelines of the National Institute of Health.
  Arms: Sleeve gastrectomy

SUMMARY:
This study aims to determine if preoperative EndoFlip measurement can effectively predict postoperative GERD-related quality of life and lower esophageal acid exposure.

DETAILED DESCRIPTION:
Enrolled patients will be subjected to a pre-operative gastroscopy, 48-Hour Bravo pH study and EndoFlip. In addition, each patient will complete a GERD-related quality of life questionnaire (GERD-HRQL scale). One year after surgery, patients will undergo a follow up a gastroscopy, pH study, EndoFlip and the same quality of life questionnaire to predict the incidence of postoperative GERD and determine the effect of sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old

Exclusion Criteria:

* Hiatal hernia > 2 cm at preoperative gastroscopy
* Erosive esophagitis at preoperative gastroscopy
* Barrett's metaplasia/dysplasia at preoperative gastroscopy
* Revision surgery before the end of the study
* Pregnancy during the study period
* Actively bleeding esophageal varices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
New-onset of gastroesophageal reflux disease | 12 months postoperatively
  total time of esophageal acid exposure (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: François-Charles Malo, Principal Investigator — Université de Sherbrooke

IPD SHARING:
Plan to Share IPD: No